CLINICAL TRIAL: NCT02141815
Title: The Effect of Arabinoxylan-oligosaccharides (AXOS) on Intestinal Generation of Microbial Metabolites in Chronic Kidney Disease
Brief Title: AXOS and Microbial Metabolites in CKD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S55578
Record Dates: First submitted 2014-05-15; First posted 2014-05-19 (Estimated); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Arabinoxylan-oligosaccharides (Experimental): Arabinoxylan-oligosaccharides 10g BID
  Interventions: Dietary Supplement: Arabinoxylan-oligosaccharides
- Maltodextrine (Placebo Comparator): Maltodextrine BID
  Interventions: Dietary Supplement: Maltodextrine

INTERVENTIONS:
Dietary Supplement: Arabinoxylan-oligosaccharides
  Other Names: AXOS
  Arms: Arabinoxylan-oligosaccharides
Dietary Supplement: Maltodextrine
  Arms: Maltodextrine

SUMMARY:
Chronic kidney disease is associated with the accumulation of various metabolites, i.e., uremic retention solutes. Evidence is mounting that the colonic microbiota contributes substantially to these uremic retention solutes. Indoxyl sulfate and p-cresyl sulfate are among the most extensively studied gut microbial metabolites, and are associated with cardiovascular disease, overall mortality and chronic kidney disease progression. The most important regulator of colonic bacterial metabolism is nutrient availability and especially the ratio of available fermentable carbohydrate to nitrogen, which can be modified by intake of so-called prebiotics (non-digestible food ingredients). Arabinoxylan oligosaccharides (AXOS) are a recently developed group of prebiotics, and already demonstrated a decreasing effect on intestinal generation of p-cresol in healthy individuals. Whether prebiotics in general, and AXOS more specifically, can influence intestinal generation of microbial metabolites in predialysis patients has not been studied to date. An interventional study with AXOS will therefore be initiated to test the hypothesis that AXOS can decrease intestinal generation and serum concentrations of microbial metabolites in patients with CKD not yet on dialysis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 85 years
* Chronic kidney disease stage 3b-4, i.e., with estimated glomerular filtration rate (CKD-epi) between 45 - 15 ml/min/m² 29
* Written informed consent

Exclusion Criteria:

* History of organic gastro-intestinal disease (e.g., inflammatory bowel disease, malignancy)
* History of colonic surgery
* Recipient of a renal or other solid organ transplant
* Use of pre-/pro-/syn- or antibiotics in preceding 4 weeks

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-05; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Serum levels of p-cresol and indole derivatives | After 4 weeks of intervention

SECONDARY OUTCOMES:
Urinary excretion rates of p-cresol and indole derivatives | After 4 weeks of intervention
Insuline resistance | After 4 weeks of intervention
  Insuline resistance, measured by HOMA index

CONTACTS AND LOCATIONS:
Overall Officials: Ruben Poesen, MD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven; Björn Meijers, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Vlaams-Brabant, Belgium

REFERENCES:
- [Derived] Cooper TE, Khalid R, Chan S, Craig JC, Hawley CM, Howell M, Johnson DW, Jaure A, Teixeira-Pinto A, Wong G. Synbiotics, prebiotics and probiotics for people with chronic kidney disease. Cochrane Database Syst Rev. 2023 Oct 23;10(10):CD013631. doi: 10.1002/14651858.CD013631.pub2. PMID 37870148
- [Derived] Poesen R, Evenepoel P, de Loor H, Delcour JA, Courtin CM, Kuypers D, Augustijns P, Verbeke K, Meijers B. The Influence of Prebiotic Arabinoxylan Oligosaccharides on Microbiota Derived Uremic Retention Solutes in Patients with Chronic Kidney Disease: A Randomized Controlled Trial. PLoS One. 2016 Apr 21;11(4):e0153893. doi: 10.1371/journal.pone.0153893. eCollection 2016. PMID 27100399